CLINICAL TRIAL: NCT07238673
Title: Dynamic Changes in Preoperative Urinary Leukocytes and Nitrite as Predictors of Infectious Complications After Percutaneous Nephrolithotomy
Brief Title: Do Dynamic Urinary Leukocyte and Nitrite Changes Improve Risk Prediction for Infectious Complications Following PCNL?
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Junhao Zheng, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GYFYZJH1015
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Kidney Calculi; Urinary Tract Infections; Sepsis
Keywords: urolithiasis; percutaneous nephrolithotomy; urinalysis; postoperative infection
MeSH Terms: conditions — Kidney Calculi; Urinary Tract Infections; Sepsis; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Percutaneous nephrolithotomy (PCNL) is widely recognized as the primary surgical approach for managing sizable and anatomically complex kidney stones., yet postoperative infection-related complications remain common and potentially severe. Preoperative urine culture plays an important role in perioperative antibiotic guidance but is limited by delayed reporting and suboptimal sensitivity. Urinalysis is simple, cost-effective, and repeatable; however, most existing studies focus on single static measurements and lack systematic evaluation of temporal trends.

Objective To evaluate the association between temporal changes in preoperative urinary white blood cells (WBC) and nitrite (NIT) and the risk of postoperative fever and urosepsis in patients undergoing PCNL.

DETAILED DESCRIPTION:
Introduction

Urolithiasis represents one of the most frequently encountered disorders in urological practice, and its global incidence has been increasing steadily in recent years, making it a significant public health concern that not only impairs patients' quality of life while creating considerable financial strain and increasing demands on healthcare systems . Percutaneous nephrolithotomy (PCNL) is now the primary therapeutic option recommended by international guidelines for medium-to-large and complex renal calculi, owing to its proven efficacy, minimal invasiveness, and rapid recovery . However, unavoidable factors during this procedure-such as high-pressure irrigation, migration of stone fragments, and injury to the renal pelvic mucosa-may facilitate the translocation of bacteria and endotoxins into the bloodstream, thereby triggering postoperative infectious complications, particularly fever and urosepsis. These complications can significantly impair postoperative recovery and prognosis and may even pose life-threatening risks .

Currently, preoperative urine culture is routinely used to assess a patient's infectious status and to guide perioperative antibiotic administration. However, this method has certain limitations, including a prolonged turnaround time (48-72 hours), susceptibility to sampling contamination, and the intermittent nature of bacteriuria, which restrict its utility in rapid clinical decision-making. In contrast, urinalysis is an economical, convenient, and repeatable test that is widely applied in preoperative evaluation. Among its parameters, urinary white blood cells (WBC) detected by microscopy and urinary nitrite (NIT) can serve as indirect indicators of urinary tract infection. Previous studies have demonstrated that preoperative WBC or NIT positivity is significantly associated with postoperative infectious complications following PCNL. A meta-analysis involving 6,113 patients reported that preoperative WBC positivity (OR ≈ 3.86) and NIT positivity (OR ≈ 7.81) were both independent risk factors. However, most of these studies were based on a single measurement and lacked a systematic evaluation of preoperative dynamic trends.

On this basis, the present study proposes a new clinical question: Can the dynamic changes in preoperative urinalysis WBC and NIT serve as effective predictors of postoperative infection risk in patients undergoing PCNL? To address this, we prospectively collected urinalysis data at admission and immediately before surgery, stratified patients according to dynamic change patterns, and analyzed the associations with postoperative fever and urosepsis, with the aim of providing a reference for clinical risk stratification and individualized anti-infective strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Renal stone diameter ≥ 2 cm, or complex renal stones, or failure of extracorporeal shock-wave lithotripsy (ESWL)
* American Society of Anesthesiologists (ASA) physical status class I or II
* Positive outpatient midstream urine culture

Exclusion Criteria:

* Age < 18 years
* Fever on admission
* Concomitant renal tumor; Active, symptomatic urinary tract infection
* Use of antibiotics for other reasons within 1 month prior to admission
* Preoperative indwelling ureteral stent, nephrostomy tube, or double-J stent
* Uncontrolled diabetes mellitus
* Chronic kidney disease stage IIIa or higher (eGFR < 60 mL/min/1.73 m²)
* Ongoing immunosuppressive therapy; Simultaneous bilateral renal stone surgery
* Severe comorbidities (e.g., respiratory or circulatory failure) that preclude anesthesia or surgery
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was based on a prospectively maintained observational cohort of patients undergoing PCNL at the Department of Urology, The First Affiliated Hospital of Guangzhou Medical University, between March 2021 and July 2025
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Fever | Within 7 days postoperatively
  Postoperative Fever was identified when body temperature reached or exceeded 38.0 °C.
Urosepsis | Within 7 days postoperatively
  Urosepsis was diagnosed according to the Sepsis-3 criteria: confirmed urinary tract infection and a Sequential Organ Failure Assessment (SOFA) score ≥ 2.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, GuangGong, China

IPD SHARING:
Plan to Share IPD: No